CLINICAL TRIAL: NCT02895685
Title: The Effect of Group Dynamics in Surgical Skill Training
Brief Title: Group Dynamics in Surgical Skill Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Copenhagen Academy for Medical Education and Simulation (Other)
Collaborators: Danish Council for Independent Research (Other); Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Diana Haunstrup Bregner Overgaard, Research Year Student, Copenhagen Academy for Medical Education and Simulation
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: KKA dyad practice
Record Dates: First submitted 2016-09-06; First posted 2016-09-12 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Technical Skills Training
Keywords: Simulation; Self-regulated training; Education; Open surgery; Dyad training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dyad training (Experimental): Participants randomized to train in pairs during the whole 6-week course
  Interventions: Other: Dyad training
- Control group: individually training (No Intervention): If randomized to train individually, participants will be instructed to do all the training individually. Participants will be instructed not to practice with others when practising at home and will only receive feedback from the expert during the expert-guided self-training. At the training at CAMES, participants will sit at separate tables.

INTERVENTIONS:
Other: Dyad training — Participants will be paired in teams at the introduction. Participants will be instructed to train and supervise each other in pairs and will receive information on how to give constructive feedback. Participants will practice in pairs during on-site classes and encouraged to train in pairs during the self-regulated training at home. At the on-site classes, participants will be instructed to practice with their partner, during the expert-guided self-training and receive all feedback in pairs. Participants will train at the same table with space for two people. Outside the classroom, participants will decide themselves when and how often they will meet to practise. Participants are instructed to actively observe his or her partner while practising and are encouraged to discuss their performance and any difficulties they encounter. Testing will be done individually. With the training log, the investigators will measure whether the participants train in pairs at home as instructed.
  Arms: Dyad training

SUMMARY:
The investigators have planned a randomized study, examining the effect of self-directed training in groups vs. individual training on trainees' acquisitions of open surgical skills.

Eighty participants who signed up for a pre-existing simulation-based course in basic open surgical skills will be randomized to practice either in pairs or individually during the course. Participants open surgical skills will be tested on a simulated skin model before and after the course. The investigators hypothesis is that dyad training will enhance self-directed learning in open surgical skills.

DETAILED DESCRIPTION:
The study is a prospective, rater-blinded, randomized, trial, examining the effect of off-site self-directed training in groups versus individual training in open surgical skills.

Setting The study will be conducted at Copenhagen Academy for Medical Education and Simulation, Rigshospitalet, Denmark. The study period will be twelve months from August 2016 to July 2017.

Basic open surgery training programme Copenhagen Academy for Medical Education and Simulation (CAMES) has developed a course in basic surgical skills in open surgery. The course is aimed at junior residents who are about to start a career in surgery. The current course is a six-week course consisting of didactic instructions with an experienced surgeon, expert-guided self-training and self-directed training at home. Each class consists of eight participants. One week before the course starts the participants meet for an introduction. At the introduction participants are provided with training material consisting of a portable knot tying and suturing kit from Ethicon, Surgical Care, Johnson and Johnson and a written material with descriptions of instruments, instructions in different technical skills and theoretical knowledge in open surgery. The following six weeks participants meet once a week for a one and a half hour on-site class in open surgical techniques. The on-site classes are held in a traditional classroom setting at CAMES and consist of didactic instructions followed by expert-guided self-training. The content of each on-site class is predefined. The participants are instructed to read the written material before the on-site classes. The first on-site classes focus on simple open surgical techniques such as knot tying and introduction to instruments and their use. The following on-site classes focuses on suturing techniques. In the end of the course, participants are introduced to more complex tasks in open surgery, such as theory in abdominal opening and closure, dissection and haemostasis (Appendix B). The participants are instructed to practice the technical skills presented in the classroom at home, using the portable knot tying and suture kit. If the participants reach a predefined level of proficiency at the examination test, held within one week after the last on-site class, they are allowed to participate in an operative course in basic open surgery techniques the following week. During the operative course basic concepts of laparotomy, ligation and dissection are practiced. The majority of the operative course focuses on practical training on sedated pigs. Groups of three trainees are supervised by an experienced surgeon.

Participants will be randomized to self-directed training at home in pairs (forty participants) or self-directed training at home individually (forty sixteen participants). All participants will follow the regular course in basic surgical skills in open surgery. Randomization will be en-bloc, so all participants following the same course, with eight participants in each course, will be randomized to follow the same instructions. Participants will be informed that they are expected to take part in classroom on-site classes, but they decide themselves when and how much time to spend practicing and which of the task presented in the classroom they practice.

Technical skill test At the introduction participant's technical skills in open surgery is assessed in a pre-test. The same test is used for examination at the end of the course (post-test). The test is composed of five basic tasks performed on a simulated skin model. The tasks are designed to explore technical skills in three different knot-tying techniques, five different suturing techniques and knowledge in selecting the right instruments and sutures. The examination instructions are presented in written format (Appendix C). Participants are given twenty-five minutes to complete the tasks. Participants are instructed to distribute their time on each task themselves. Unlimited time is given before the test starts to read the instructions carefully and to select the sutures needed. Tests are recorded on video. The camera is placed so only the hands of the trainee and the operation field is showed on the video. Audio will be deleted to allow for blinded rating. To pass the course, the trainees must achieve a predefined proficiency level corresponding to fifty percent (15 points) of the maximum score (30 point) at the post-test. The test will be performed at CAMES assuring optimal height and light setting at every test session.

Task 1: The participant is instructed to close a five cm wound using far-far near-near running suturing technique, 3-0 monofilament, nonabsorbable suture, anatomical forceps, and to start and end the suture using two hand knot tying technique.

Task 2: The participant is instructed to close a five cm wound, the skin model simulates the fascia, they are asked to use an absorbable suture, De Bakey forceps and one hand knot tying technique to start and end the suturing.

Task 3: The participant is instructed to close a five cm wound using subcuticular suturing technique, a 4-0 absorbable suture, anatomical forceps, and to start and end the suture using instrumental knot tying technique.

Task 4: The participant is instructed to demonstrate three far-far near-near interrupted sutures on a five cm wound, using 4-0 monofilament, nonabsorbable suture, anatomical forceps and to close each suture with one hand knot tying technique.

Task 5: The participant is instructed to close a five cm wound using simple interrupted suturing technique. The participant decides themselves which suture, instruments and knot tying technique they will use.

Participants are instructed to show what kind of sutures that have chosen for each task to the camera.

Training log Participants will be asked to keep a training log with details of time spend on training and number of training sessions. The training log will contain information on which type of task is practised and if the training is performed in pairs. Also time spend in the operation room, assisting or performing open surgery will be registered (APPENDIX D). Every week when the participants meet for the on-site class held at CAMES, the training log will be copied, to ensure the participants fill in the training log correctly and regularly.

Expert assessment Two experts in surgery will do the ratings based on video-recordings. One rater will be blinded for both the randomization (dyad-training versus individually training) and who is performing on the video-recording. The other rater will teach the on-site classes and rate the examination tests, and is therefore not blinded for the randomization for the post-test. However, this rater will still be blinded for the randomization for the pre-test ratings and who that perform on the video-recording. The Objective Structured Assessment of Technical Skills (OSATS) is used as the primary endpoint of this study. OSATS is a validated assessment tool for the evaluation of general surgical skills[15, 16]. OSATS consists of a five-point global rating scale (GRS) and task specific checklists[15]. Only the GRS will be used for assessment, as no full procedures are performed in the test. A modified GRS will be used, as the audio will be deleted from all videos and no assistant will be available during testing. Using the modified GRS trainees will be evaluated on the following categories: 1) respect for tissue, 2) time and motion, 3) instrument handling, 4) knowledge of instruments, 5) flow of operation and forward planning and 6) knowledge of specific procedure (Appendix E).

Handling of adverse events during testing

During testing there is a risk of adverse events. They should be handled as follows:

The practical equipment fails:

Testing is stopped. If equipment fail is repairable on the testing session, testing is restarted at the point it was stopped. If not, the testing session is seen as failed and the testing session will not be used or counted as an attempt. A new test will be performed.

The simulated skin model becomes detached from the table:

The participant is allowed to fix the simulated skin model to the table and will continue to finish the task. If this is not possible, a score of zero will be given.

Other interruptions during testing:

Testing is stopped. If the interruption can be overcome during the testing session, testing is restarted at the point it was stopped. If not, the testing session is seen as a failed testing session and will not be used.

A test session which fails due to adverse events will not be used in the final analysis and a new test session will be arranged.

Study participants Participants are medical doctors with a surgical interest and medical students in relevant jobs related to surgery (internships, research year) participating in the course in basic surgical skills in open surgery. Eighty trainees', who sign up for the current course in basic open surgical skills, will be enrolled in the study.

Note:

Base-line testing (pre-test) for 15 participants have been carried out in august 2016. These participants where randomized according to the protocol. No changes has been made to the protocol, and data has not been analyzed, since no post-testing has been carried out. The data from the first 15 participants will not be obtained and analyzed before the post-test at the end of september.

ELIGIBILITY:
Inclusion Criteria:

* The participants may enter the study if any of the following apply:

Medical doctor from a department in the Capital Region and the region of Zeeland in Denmark.

* Medical students employed in internships or research year in surgical departments in the Capital Region and the region of Zeeland in Denmark.
* The participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* The participants may not enter the study if any of the following apply:
* The participant have performed more than 50 open surgical procedures.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
To examine the effect of off-site self-directed training in groups vs. individual training | 12 months
  Differences between pre-test and post-test scores in basic tasks on a simulated model

SECONDARY OUTCOMES:
To examine the effect of off-site self-directed training in groups vs. individual training | 12 months
  Differences in time(mins.) spend on self-directed training
To examine the effect of off-site self-directed training in groups vs. individual training | 12 months
  Differences in number of self-directed training sessions
To examine the effect of off-site self-directed training in groups vs. individual training | 12 months
  Differences in number of dyadic training sessions at home
To examine the effect of off-site self-directed training in groups vs. individual training | 12 months
  Differences in number of participants completing the course
To examine the effect of off-site self-directed training in groups vs. individual training | 12 months
  Differences in attendance in on-site classes
To examine the effect of off-site self-directed training in groups vs. individual training | 12 months
  Differences in number of tasks performed per trainee during self-directed training (hands-on time)
To examine the effect of off-site self-directed training in groups vs. individual training | 12 months
  Differences in rating scores (blinded, non-blinded)

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen Academy for Medical Education and Simulation, Copenhagen, Copenhagen Ø, Denmark

IPD SHARING:
Plan to Share IPD: No